CLINICAL TRIAL: NCT05220072
Title: An Open Label, Single-dose, Single-period Study Designed to Assess the Mass Balance Recovery, Metabolite Profile and Metabolite Identification of Carbon-14 BIA 28-6156 in Healthy Male Subjects
Brief Title: Mass Balance Recovery and Metabolite Identification of Carbon-14 BIA 28-6156
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bial R&D Investments, S.A. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BIA 28-6156-106
Record Dates: First submitted 2021-11-18; First posted 2022-02-02 (Actual); Last update posted 2025-05-28 (Actual); Status verified 2025-05

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Carbon-14 BIA 28-6156 (Experimental): Healthy volunteers receive a single dose of Carbon-14 BIA 28-6156
  Interventions: Drug: Carbon-14 BIA 28-6156

INTERVENTIONS:
Drug: Carbon-14 BIA 28-6156 — Carbon-14 BIA 28-6156 60 mg, containing NMT 3.7 MBq Carbon-14

SUMMARY:
The study is designed to determine the absorption, distribution, metabolism and elimination (ADME) of BIA 28-6156 in humans, further explore the PK of BIA 28-6156, evaluate the extent of distribution of total radioactivity into blood cells, provide additional safety and tolerability information and collect samples for metabolite profiling and structural identification.

DETAILED DESCRIPTION:
This is an open-label, single-dose, single period study in healthy male subjects. It is planned to enroll 6 subjects. All subjects will receive a single oral dose Carbon-14 BIA 28-6156. Blood samples will be collected at regular intervals for PK analysis, mass balance and metabolite profiling and identification from pre-dose up to 240 h post-dose. Urine and faecal samples will be collected at regular intervals for mass balance and metabolite profiling and identification from pre-dose until the mass balance criteria have been met.

ELIGIBILITY:
Inclusion Criteria:

* Healthy males aged 30 to 65 years inclusive
* Body mass index (BMI) of 18.0 to 35.0 kg/m2
* Must be willing and able to communicate and participate in the whole study
* Must have regular bowel movements
* Must provide written informed consent
* Must agree to adhere to contraception requirements

Exclusion Criteria:

* Subjects who have received any IMP in a clinical research study within the 90 days prior to Day 1
* Subjects who are, or are immediate family members of, a study site or sponsor employee
* Evidence of current SARS-CoV-2 infection from results of diagnostic tests or from symptoms reported at screening or admission
* History of any drug or alcohol abuse in the past 2 years
* Regular alcohol consumption
* A confirmed positive alcohol breath test at screening or admission
* Current smokers and those who have smoked within the last 12 months.
* Current users of e-cigarettes and nicotine replacement products and those who have used these products within the last 12 months
* Subjects with pregnant or lactating partners
* Radiation exposure, including that from the present study, excluding background radiation but including diagnostic x-rays and other medical exposures, exceeding 5 mSv in the last 12 months or 10 mSv in the last 5 years.
* Subjects who do not have suitable veins for multiple venepunctures/cannulation
* Clinically significant abnormal clinical chemistry, haematology or urinalysis. Subjects with Gilbert's Syndrome are allowed.
* Confirmed positive drugs of abuse test result
* Positive hepatitis B surface antigen (HBsAg), hepatitis C virus antibody (HCV Ab) or human immunodeficiency virus (HIV) antibody results
* Evidence of renal impairment at screening, as indicated by an estimated creatinine clearance (CLcr) of <80 mL/min using the Cockcroft-Gault equation
* History of clinically significant cardiovascular, renal, hepatic, dermatological, chronic respiratory or gastrointestinal disease, neurological or psychiatric disorder
* Serious adverse reaction or serious hypersensitivity to any drug or the formulation excipients
* Presence or history of clinically significant allergy requiring treatment. Hay fever is allowed unless it is active
* Donation of blood or plasma within the previous 3 months or loss of greater than 400 mL of blood
* Subjects who are taking, or have taken, any prescribed or over-the-counter drug or herbal remedies (other than up to 4 g of paracetamol per day) in the 14 days before IMP administration.
* Failure to satisfy the investigator of fitness to participate for any other reason

Ages: 30 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2021-08-28 (Actual); Primary Completion 2021-10-16 (Actual); Study Completion 2021-10-16 (Actual)

PRIMARY OUTCOMES:
Mass balance recovery of total radioactivity in all excreta (urine and faeces) | Urine: Day 1 through Day 11, Faeces: Day -1 through Day 11
  CumAe and Cum%Ae
Collection of urine and faecal samples for total radioactivity | Urine and Faeces: Pre-dose until 288 hours post-dose
  Total radioactivity for total recovery of Carbon-14 BIA28-6156
Collection of plasma samples for metabolite profiling | Pre-dose until 240 hours post-dose
  Collection of major metabolites for metabolite profiling of BIA28-6156
Collection of plasma samples for structural identification | Pre-dose until 240 hours post-dose
  Identification of chemical structure of major metabolites of BIA28-6156
Collection of whole blood samples for total radioactivity | Pre-dose until 240 hours post-dose
  Total radioactivity for total recovery of Carbon-14 BIA28-6156

SECONDARY OUTCOMES:
Determination of routes and rates of elimination of Carbon-14 BIA 28-6156 | Day 1 through Day 11
Identification of the chemical structure of each metabolite accounting for more than 10% by AUC of circulating plasma total radioactivity and more than 10% of total radioactive dose | Urine and Faeces: Day 1 through Day 11, Plasma: Day 1 through Day 7
Measurement of BIA 28-6156 PK parameters | Day 1 through Day 11
Evaluation of whole blood: plasma concentration ratios for total radioactivity | Day 1 through Day 7
Adverse events (AEs) | Screening through Day 11

CONTACTS AND LOCATIONS:
Overall Officials: Somasekhara Menakuru, MBBS,MS,MRCS,DPM,MFPM, Principal Investigator — Quotient Sciences
Locations (1):
- Quotient Sciences, Ruddington, Nottingham, United Kingdom

IPD SHARING:
Plan to Share IPD: No